CLINICAL TRIAL: NCT03300999
Title: The Effects of Daily Ginger Tea Consumption in Reducing Discomfort During Menstruation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5170302
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Discomfort
Keywords: ginger tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginger Tea (Experimental): * End of the second menstruation cycle - Start of the third menstruation cycle: Subjects will take ginger tea daily, avoid home remedies, refrain from taking pain medications and supplements, and keep track of ginger tea intake by placing a check mark each day in the daily log checklist.
  * Start of the third menstruation cycle - End of the third menstruation cycle: Subjects will drink ginger tea daily. Subjects will rate discomfort using the visual analog pain scales and the symptom checklist at the end of each day during menstruation.
  * After the third menstruation cycle ends: Subjects will meet with student investigators at a location convenient to the subject to turn in daily logs, visual analog pain scales, and symptom checklists.
  Interventions: Dietary Supplement: ginger tea
- No Ginger Tea (No Intervention): * End of the first menstruation cycle - Start of the second menstruation cycle: Subjects will not take ginger tea, avoid home remedies, and refrain from taking pain medications or supplements.
  * Start of the second menstruation cycle - End of the second menstruation cycle: Subjects will rate discomfort using the visual analog pain scales and symptom checklist during menstruation. Subjects will meet with student investigators at a convenient location to the subject and will complete surveys and questionnaires. Subjects will be given daily logs, visual analog pain scales, symptom checklists, and supplies for the ginger tea.

INTERVENTIONS:
Dietary Supplement: ginger tea — 1. Ginger tea - Swanson Organic: 100% Certified Organic Ginger Root Tea
  • Subjects will use one tea bag (contains two grams ginger root), mix with eight ounces of boiling water, steep for three minutes, and allow it to cool to room temperature before drinking. This will be done every day for one month before their third menstruation cycle and during their third menstruation cycle.
  Arms: Ginger Tea

SUMMARY:
The purpose of our graduate student research study is to observe the effect of drinking ginger tea daily on period discomfort.

DETAILED DESCRIPTION:
* Day 1: Subjects will sign informed consent and will go over the introduction, purpose, procedures, and compliance with student investigators. Subjects will then be given a sample of ginger tea that will be used for the study and will be asked if they think they can drink this daily for a month. They will also be asked if they have regular menstrual cycles and agree to stop home remedies and stop taking pain medications or herbal supplements for a period of three menstruation cycles.
* Start/During the first menstruation cycle: Subjects will meet with student investigators at a convenient location to the subject and will complete surveys and questionnaires. Subjects will be given visual analog pain scales and symptom checklists that need to be completed during their second menstruation cycle.
* End of the first menstruation cycle - Start of the second menstruation cycle: Subjects will not take ginger tea, avoid home remedies, and refrain from taking pain medications or supplements.
* Start of the second menstruation cycle - End of the second menstruation cycle: Subjects will rate discomfort using the visual analog pain scales and symptom checklist during menstruation. Subjects will meet with student investigators at a convenient location to the subject and will complete surveys and questionnaires. Subjects will be given daily logs, visual analog pain scales, symptom checklists, and supplies for the ginger tea.
* End of the second menstruation cycle - Start of the third menstruation cycle: Subjects will take ginger tea daily, avoid home remedies, refrain from taking pain medications and supplements, and keep track of ginger tea intake by placing a check mark each day in the daily log checklist.
* Start of the third menstruation cycle - End of the third menstruation cycle: Subjects will rate discomfort using the visual analog pains scales and symptom checklist during menstruation.
* After the third menstruation cycle ends: Subjects will meet with student investigators at a location convenient to the subject to turn in daily logs, visual analog pain scales, and symptom checklists.

ELIGIBILITY:
Inclusion Criteria:

1. female within age range
2. regular menstrual cycles
3. experiencing period cramps
4. agrees to refrain from taking any pain medications, herbal supplements, or use home remedies such as heating pads that are known to alleviate menstrual cramps during the study period
5. after sampling the ginger tea, the subject must agree to drink ginger tea daily.

Exclusion Criteria:

1. women who take oral contraceptives
2. work night shifts
3. allergic to ginger
4. lactating
5. female-related uterine problems such as fibroids and polycystic ovarian syndrome who suffer from secondary dysmenorrhea

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female with regular menstrual cycles
Enrollment: 15 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | Change between Day 1 of the Second Menstruation Cycle and Day 28 of the Second Menstruation Cycle. Cycle is 28 days.
  • The Visual Analogue scale is a form of a Likert scale that gives the interviewee maximum freedom to estimate their pain intensity. The interviewee will mark a line along the 10-cm scale which they perceive corresponds best to their exact pain intensity every day for the duration of the study. A score of zero indicated no pain and a score of 10 indicated the most severe pain felt.
Visual Analog Pain Scale | Change between Day 1 of the Third Menstruation Cycle and Day 28 of the Third Menstruation Cycle. Cycle is 28 days.
  • The Visual Analogue scale is a form of a Likert scale that gives the interviewee maximum freedom to estimate their pain intensity. The interviewee will mark a line along the 10-cm scale which they perceive corresponds best to their exact pain intensity every day for the duration of the study. A score of zero indicated no pain and a score of 10 indicated the most severe pain felt.

SECONDARY OUTCOMES:
SF-36 Quality of Life Survey | On any day between Day 1 and Day 28 of the first menstruation cycle. Cycle is 28 days.
  RAND developed this validated survey and it is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. This survey consists of eight scaled scores which are the weighted sums of the questions in each section. The sections include vitality, physical functioning, bodily pain, physical role functioning, general health perception, emotional role functioning, social role functioning, and mental health. Each scale is transformed into a 0-100 scale and the lower score indicates more disability while the higher represents less disability. It can take participants at least half an hour to complete and will be assessed over a one-month period.
SF-36 Quality of Life Survey | Day 28 of the second menstruation cycle. Cycle is 28 days.
  RAND developed this validated survey and it is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. This survey consists of eight scaled scores which are the weighted sums of the questions in each section. The sections include vitality, physical functioning, bodily pain, physical role functioning, general health perception, emotional role functioning, social role functioning, and mental health. Each scale is transformed into a 0-100 scale and the lower score indicates more disability while the higher represents less disability. It can take participants at least half an hour to complete and will be assessed over a one-month period.
SF-36 Quality of Life Survey | Day 28 of the third menstruation cycle. Cycle is 28 days.
  RAND developed this validated survey and it is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. This survey consists of eight scaled scores which are the weighted sums of the questions in each section. The sections include vitality, physical functioning, bodily pain, physical role functioning, general health perception, emotional role functioning, social role functioning, and mental health. Each scale is transformed into a 0-100 scale and the lower score indicates more disability while the higher represents less disability. It can take participants at least half an hour to complete and will be assessed over a one-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Kyndra Woosley, MS RD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No